CLINICAL TRIAL: NCT04306939
Title: Genomic Resources for Enhancing Available Therapies (GREAT1.0) Study
Acronym: GREAT1
Status: Suspended | Type: Observational
Why Stopped: Suspended for analysis and to consider further enrollment.
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, David Binion, MD, Professor, University of Pittsburgh
Other Study IDs: STUDY19020035
Record Dates: First submitted 2019-12-16; First posted 2020-03-13 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pancreatitis; Inflammatory Bowel Diseases; Hepatitis; NASH - Nonalcoholic Steatohepatitis; Acute Pancreatitis; Rheumatoid Arthritis; Diabetes Mellitus; Dyslipidemias; Multiple Sclerosis; Irritable Bowel Syndrome; Chronic Pain; Chronic Disease; Chronic Kidney Diseases; Crohn Disease; Celiac Disease; Biliary Cirrhosis; Bile Acid Synthesis Defect; Gastritis; Cholecystitis; Cholelithiases; IPMN; Cyst Pancreas; Cystic Fibrosis; Pancreatic Exocrine Insufficiency; Diarrhea Chronic; Constipation - Functional; Constipation Chronic Idiopathic
Keywords: fibrosis; chronic inflammation
MeSH Terms: conditions — Pancreatitis, Chronic; Inflammatory Bowel Diseases; Hepatitis; Non-alcoholic Fatty Liver Disease; Pancreatitis; Arthritis, Rheumatoid; Diabetes Mellitus; Dyslipidemias; Multiple Sclerosis; Irritable Bowel Syndrome; Chronic Pain; Chronic Disease; Renal Insufficiency, Chronic; Crohn Disease; Celiac Disease; Liver Cirrhosis, Biliary; Gastritis; Cholecystitis; Cholelithiasis; Pancreatic Cyst; Cystic Fibrosis; Exocrine Pancreatic Insufficiency; Fibrosis | interventions — Phlebotomy; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples will provide functional and mechanistic information about subject health, disease or state.
  The protocol allows the collection of biological waste, defined as any biological sample that is left over from a laboratory test or procedure such as surgery or endoscopy.
  Blood sample in addition to waste may be obtained at the time of venipuncture for clinical testing to optimize sample collection for biomarkers that may be affected by delays in clinical testing. An extra 21cc of blood can be accepted, up to 4 time a year, and with the approval of the attending physician Research blood collection is also an option via venipuncture if the subject is not scheduled for clinical testing. This will also be limited to 21cc of blood, up to 4 time a year, and with the approval of the attending physician.
  Research samples that are non-invasive, such as those from saliva, urine, stool, hair, etc. may also be collected with patient consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case/Chronic complex disorders: Chronic complex disorders are composed of multiple population sub classifications - many of which have not been fully defined. Thus, all eligible patients should be included to maximize study power. Sufficient numbers of controls, those individuals in the general population, who may or may not have complex disorders are needed to match future comparison studies for a subset of questions, and so should also be included.
  Interventions: Other: venipuncture; Behavioral: Questionnaires; Other: Additional Sample Collections
- Control: The number of controls that are anticipated for this study is less than patient numbers since they will not be needed for calculating the minor allele frequency of the majority of genetic polymorphism of interest in genetic association studies. This data is already available in public and research databases. Controls will be useful for evaluating case report form questions, providing assessment of the local genetic pool, and for possibly participating in future studies as provided by the consent.
  Interventions: Other: venipuncture; Behavioral: Questionnaires; Other: Additional Sample Collections

INTERVENTIONS:
Other: venipuncture — Research blood collection is also an option via venipuncture if the subject is not scheduled for clinical testing. This will also be limited to 21cc of blood, up to 4 time a year, and with the approval of the attending physician.
Behavioral: Questionnaires — PROMIS-43 Profile, PROMIS-29 Profile, Global Health Scale and Hospital Anxiety and Depression Scale (HADS). Additional assessments can be approved and administered per specific disease sub-category.
Other: Additional Sample Collections — We may also contact subjects to request additional blood, saliva, cheek swab, hair, urine, or stool with their permission. This will be limited to no more than 4 teaspoons of blood and will happen no more than 4 times per year.

SUMMARY:
This is a prospective, descriptive, observational research study designed to observe and document the clinical practice by domain experts, and how the knowledge of new findings that are published in the medical literature affect clinical decision making.

The study will evaluate risk factors and co-variants, including genetic variants that are associated with disease progression such as pain, inflammation, organ dysfunction, disability and quality of life.

DETAILED DESCRIPTION:
The Genomic Resource to Enhance Available Therapies (GREAT1.0) Study is a research program for personalized medicine. It is a highly annotated genetic and biosample resource for multiple nested observational cohort studies. It is designed to begin to understand the mechanisms underlying complex diseases using clinical information from the UPMC electronic health record (EHR), from case-report forms, and from biological samples.

Aim 1. To test the hypothesis that point-of-care electronic health record (EHR)-based phenotyping and clinical measures will be useful for classifying patient by disease risk, subtype, activity, complications, quality of life or using statistical or systems approaches.

Aim 2. To test the hypothesis that common diseases can be subtyped using genotype data.

Aim 3. To test the hypothesis biological samples will provide additional functional and mechanistic information about subject health, disease or state.

The study will be conducted using UPMC patients and population controls. Consent will allow EHR and/or case report form data, plus biological samples to be given a unique code number and transferred to researchers for analysis. Consent will also allow for a secure link to be maintained allowing the research data or samples to be updated, and to contact the clinical team and/or subject to provide them with additional information.

ELIGIBILITY:
Inclusion Criteria:

Case Subjects

* Clinical diagnosis of a chronic disease or disorder (ex. pancreatitis, hepatitis or fatty liver, inflammatory bowel disease, irritable bowel syndrome, diarrhea, constipation, chronic pain syndromes, diabetes, hypertension, cardiovascular disease, chronic kidney disease, chronic neurologic disorders, rheumatological disorders, endocrine disorders, chronic pulmonary diseases, sinorespiratory disorders, chronic skin diseases, cancers and related disorders)
* Ability to read and write in English;
* Ability to provide informed consent

Control Subjects

• UPMC patients age 12 years without a chronic disorder.

Exclusion Criteria:

* Chronic infectious disease as the primary medical problem
* Less than 12 years of age
* Inability of the subject to understand the protocol
* Inability to the subject provide informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen in a UPMC facility with available electronic health records
Sampling Method: Non-Probability Sample
Enrollment: 120000 (Estimated)
Dates: Start 2014-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Define the molecular disorders contributing to clinicopathological disease definitions for common complex disorders | through study completion, an average of 1 year
  Diseases are defined by symptoms and pathologic features in specific tissues. The study uses genetic variants associated with disease to define the underlying genes associated with disease, and uses cell biology methods to understand which mechanisms within the specialized cells lead to disease under specific conditions.
Define risk factors for disease progression, severity, complications and poor quality of life. | through study completion, an average of 1 year
  Life-style (e.g. alcohol, smoking, diet, exercise), medications, metabolic, genetic and epigenetic factors alter the features of disease. Nested studies, subgroup analysis, stepwise regression, statistical and machine learning will be used to develop disease models where early intervention may alter disease progression and severity.
Common disease mechanisms and repurposing of medications. | through study completion, an average of 1 year
  Many chronic diseases, including inflammatory and autoimmune diseases, have similar disease features that arise in different organs. Harmonization of similar disease processes in different organs will be used to increase study power, and to determine if there is evidence that therapeutic interventions for one disease may be effective in another disease, providing evidences to consider drug repurposing and new treatment approaches.

SECONDARY OUTCOMES:
Pain profile | through study completion, an average of 1 year
  Pain is measured using visual analogue scales, pain quality, pattern and interference using standardized questionnaires. Patients with similar disease stages and severity often have markedly different levels of pain. Validated tools will be used to observe responses to disease treatments between similar patients, and to observe factors that may be targetable to lessen pain in future intervention studies.
Patient Reported Global Health Assessment | through study completion, an average of 1 year
  PROMIS29 It is a comprehensive measure in that it is assessing multiple aspects of mental, physical, and social health.

CONTACTS AND LOCATIONS:
Overall Officials: David C Binion, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whitcomb DC. Primer on Precision Medicine for Complex Chronic Disorders. Clin Transl Gastroenterol. 2019 Jul;10(7):e00067. doi: 10.14309/ctg.0000000000000067. PMID 31335357